CLINICAL TRIAL: NCT02281331
Title: Evaluation of the Effects of a Combined Resistance and High-intensity Interval Exercise Training Program, Along With Nutritional Supplementation, on Strength and Physical Function in Older Men
Brief Title: Optimal Exercise Training and Nutrition Supplementation in Older Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REB 14-677
Record Dates: First submitted 2014-10-08; First posted 2014-11-03 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Aging
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supplement (Active Comparator): Each day, participants in this group will receive a supplement that provides a total of protein, creatine monohydrate, calcium, vitamin D and carbohydrate. This supplement will be provided to participants in beverage format, twice daily.
  Interventions: Dietary Supplement: Supplement
- Placebo (Placebo Comparator): The placebo will provide participants with maltodextrin (carbohydrate) and sucrose.
  Interventions: Dietary Supplement: Supplement

INTERVENTIONS:
Dietary Supplement: Supplement — supplement/placebo plus exercise training

SUMMARY:
As we age we tend to lose muscle mass and strength. These losses contribute to the increased incidence of falls and fractures, metabolic diseases such as type 2 diabetes, loss of independence and reduced quality of life in the elderly. As the number of seniors increases worldwide, it is becoming more and more important to develop strategies to counteract this loss of muscle mass and strength, and promote healthy aging. Fortunately, relatively simple lifestyle modifications are the most potent defense strategies. Exercises such as weight lifting and high-intensity interval exercise (HIIT), which consists of short, repeated bouts of vigorous aerobic exercise interspersed with period of rest, are the most effective in promoting gains in muscle mass and strength. Additionally, components of foods like whey (a protein found in milk), creatine (found in meat), calcium and vitamin D have been shown to independently increase strength. In this study, we are looking to determine how much we can increase muscle strength in older men who are put on an 12 week exercise training program that combines weight lifting and HIIT, and who consume a daily supplement that contains whey protein, creatine, calcium and vitamin D.

DETAILED DESCRIPTION:
Please see other documentation.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary (no participation in a structured exercise training program in past 6 months)
* BMI between 18.5-30.0 kg/m2
* Weight stable for past 6 months
* Normal resting blood pressure, or stage I hypertension

Exclusion Criteria:

* Smoking
* Use of simvastatin or atorvastatin
* Use of non-steroidal anti-inflammatory drugs
* Injuries that prevent safe-participation in an exercise training program
* Prescription blood thinners
* Diabetes or other metabolic disorders
* Cardiac or gastro-intestinal problems
* Infectious disease or cancer

Min Age: 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Muscle mass | 12 weeks
  DXA, ultrasound

SECONDARY OUTCOMES:
Muscle protein synthesis | 12 weeks
  The incorporation of a stable isotope (deuterium) into muscle tissue will allow for the determination of fractional synthetic rate, which is indicative of muscle protein synthesis.
Satellite cell number, density, type I/type II fibre specific satellite cells and myonuclear domain | 12 weeks
  Histochemical methods will be used to determine how the supplement and training affect muscle growth and regenerative capacity, specifically the behaviour of satellite cells.
Glycemic control | 12 weeks
  Oral glucose tolerance test
Cognitive function | 12 weeks
  Questionnaires and simple computer-based identification, reaction time and memory tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Phillips, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster Univeristy, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Bell KE, Fang H, Snijders T, Allison DJ, Zulyniak MA, Chabowski A, Parise G, Phillips SM, Heisz JJ. A Multi-Ingredient Nutritional Supplement in Combination With Resistance Exercise and High-Intensity Interval Training Improves Cognitive Function and Increases N-3 Index in Healthy Older Men: A Randomized Controlled Trial. Front Aging Neurosci. 2019 May 9;11:107. doi: 10.3389/fnagi.2019.00107. eCollection 2019. PMID 31143111
- [Derived] Bell KE, Brook MS, Snijders T, Kumbhare D, Parise G, Smith K, Atherton PJ, Phillips SM. Integrated Myofibrillar Protein Synthesis in Recovery From Unaccustomed and Accustomed Resistance Exercise With and Without Multi-ingredient Supplementation in Overweight Older Men. Front Nutr. 2019 Apr 11;6:40. doi: 10.3389/fnut.2019.00040. eCollection 2019. PMID 31032258
- [Derived] Snijders T, Bell KE, Nederveen JP, Saddler NI, Mazara N, Kumbhare DA, Phillips SM, Parise G. Ingestion of a Multi-Ingredient Supplement Does Not Alter Exercise-Induced Satellite Cell Responses in Older Men. J Nutr. 2018 Jun 1;148(6):891-899. doi: 10.1093/jn/nxy063. PMID 29878269
- [Derived] Bell KE, Snijders T, Zulyniak M, Kumbhare D, Parise G, Chabowski A, Phillips SM. A whey protein-based multi-ingredient nutritional supplement stimulates gains in lean body mass and strength in healthy older men: A randomized controlled trial. PLoS One. 2017 Jul 18;12(7):e0181387. doi: 10.1371/journal.pone.0181387. eCollection 2017. PMID 28719669